CLINICAL TRIAL: NCT03153865
Title: New Therapeutic System of Unruptured Intracranial Aneurysms Based on Big Data From Chinese Population
Acronym: NATIONAL-1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Qinghai Huang, Principal Investigator, Changhai Hospital
Other Study IDs: CHEC2017-073
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Unruptured Cerebral Aneurysm; Treatment Strategy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, multicenter, observational study, aiming at comparing the Safety and effectiveness among the different surgical treatment of unruptured intracranial aneurysms in China, so as to improve the diagnosis and treatment of unruptured intracranial aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with unruptured intracranial saccular aneurysm on CTA, MRA or DSA.
* patients willing to participate in this clinical trial and attach to regular follow up.

Exclusion Criteria:

* intracranial aneurysm correlating to AVM.
* intracranial non-saccular aneurysm.
* the rupture or unrpture of the aneurysm confirmed on CTA、MRA or DSA.
* patients unwilling to participate in this clinical trial and attach to regular follow up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients diagnosed with unruptured intracranial saccular aneurysm at all age.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-06-02 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
mortality and disability | through study completion, an average of 1 year
  the rate of death and disable

SECONDARY OUTCOMES:
recurrence rate | 1 month, 6 months and 1 year after surgery;
progression of disease | 1 month, 6 months and 1 year after conservative treatment；
  enlarge or ruptured of the aneurysm

OTHER OUTCOMES:
the level of psychological states changes | 1 month, 6 months and 1 year after been aware of the disease
  The Sheet for Affective Disorders was used to record the level of psychological states changes in every participant when they were aware of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Qinghai Huang, MD, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No